CLINICAL TRIAL: NCT03462251
Title: A Randomized, Open-label, Multicenter, Two-arm, Phase III Study to Evaluate Efficacy and Quality of Life in Patients With Metastatic Hormone Receptor-positive HER2-negative Breast Cancer Receiving Ribociclib in Combination With Endocrine Therapy or Chemotherapy With or Without Bevacizumab in First Line
Brief Title: Ribociclib and Endocrine Therapy or Chemotherapy With or Without Bevacizumab for Metastatic Breast Cancer in First Line
Acronym: RIBBIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: iOMEDICO AG (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOM-050371
Record Dates: First submitted 2018-02-16; First posted 2018-03-12 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Hormone Receptor Positive Tumor; HER 2 Negative Breast Cancer
Keywords: Breast Cancer; HR positive; HER2 negative; Mamma carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Aromatase Inhibitors; Fulvestrant; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Combination of ribociclib and aromatase inhibitor or fulvestrant
  Interventions: Combination Product: Ribociclib and aromatase inhibitor or fulvestrant
- Arm B (Active Comparator): Capecitabine + bevacizumab OR Paclitaxel +/- bevacizumab
  Interventions: Combination Product: Capecitabine + bevacizumab OR Paclitaxel +/- bevacizumab

INTERVENTIONS:
Combination Product: Ribociclib and aromatase inhibitor or fulvestrant — Combination of ribociclib and aromatase inhibitor or fulvestrant
  Arms: Arm A
Combination Product: Capecitabine + bevacizumab OR Paclitaxel +/- bevacizumab — Capecitabine with bevacizumab OR Paclitaxel with or without bevacizumab
  Arms: Arm B

SUMMARY:
This study is designed to evaluate the efficacy and safety of first-line treatment ribociclib in combination with aromatase inhibitor (AI) or fulvestrant OR capecitabine with bevacizumab OR paclitaxel with / without bevacizumab in patients with HR-positive, HER2-negative advanced breast cancer with visceral metastasis.

Half of the patients will receive a combination of ribociclib and AI/fulvestrant while the other half will receive capecitabine + bevacizumab or paclitaxel +/- bevacizumab.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, two-arm, multicenter, interventional phase III trial in Germany. The study will include adult women with HR-positive, HER2-negative advanced breast cancer with visceral metastases, who received no prior therapy for advanced disease.

158 patients will be enrolled and randomized 1:1 (stratified by the presence of lung and / or liver metastases) to receive Arm A: a combination of ribociclib and AI or fulvestrant; OR Arm B: capecitabine + bevacizumab OR paclitaxel +/- bevacizumab

Treatment will be continued until disease progression, intolerable toxicity or death. Progression-free survival (PFS) will be based on tumor assessments by local radiologists/investigator using RECIST v1.1 criteria. Treatment might be continued beyond RECIST-defined progressive disease (PD) in case of negligible or clinically irrelevant disease progression according to the investigator's discretion until clinically relevant disease progression or symptomatic deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Any menopausal status. If pre-/perimenopausal, agreement to receive LHRH agonist (goserelin or leuprorelin) / ovarian ablation in case of randomization to arm A
* Locally confirmed diagnosis of metastatic adenocarcinoma of the breast without prior systemic antineoplastic therapy in the palliative setting.
* Hormone receptor (HR)-positive disease, defined as estrogen receptor (ER)-positive and/or progesterone receptor (PgR)-positive.
* Human epidermal growth factor receptor 2 (HER2)-negative disease (defined as immunohistochemistry (IHC) status HER2 negative/+ or IHC HER2++ with chromosomal in situ hybridization (CISH)/fluorescent in situ hybridization (FISH) negative).
* Presence of visceral metastases (additional non-visceral metastases are allowed).
* Presence of target and / or non-target lesions according to RECIST v1.1
* Patients eligible for palliative treatment with AI / fulvestrant + ribociclib and capecitabine + bevacizumab or paclitaxel + / - bevacizumab according to the respective SmPCs.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Adequate organ and bone marrow function within 7 days prior to randomization.
* Standard 12-lead ECG values: QT Interval Corrected by the Fridericia Correction Formula (QTcF) interval at screening < 450 msec; Mean resting heart rate 50-90 bpm (determined from the ECG)
* Signed written informed consent prior to beginning of protocol-specific procedures.

Exclusion Criteria:

* Any prior systemic palliative therapy
* Prior treatment with any cyclin-dependent kinase 4/6 (CDK4/6) inhibitor.
* Prior adjuvant or neoadjuvant taxane therapy if last application within 12 months prior to entering the study.
* Patient is concurrently using other anti-cancer therapy.
* Patient has had major surgery within 28 days prior to randomization or has not recovered from major side effects or wound is not fully recovered.
* Patient has received extended-field radiotherapy ≤ 4 weeks or limited-field radiotherapy ≤ 2 weeks prior to randomization.
* Known hypersensitivity to ribociclib, AI, paclitaxel, bevacizumab or any of their excipients, or against peanut, soya, Chinese hamster ovarian cell products or macrogolglycerol ricinoleate-35.
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality (e.g. history of myocardial infarction within 6 months prior study entry, long QT syndrome, clinically significant cardiac arrhythmias or systolic blood pressure > 140 or < 90 mmHg or diastolic blood pressure > 90 mmHg).
* Patient has history of arterial thrombosis within 12 months prior to entering the study.
* Patient has proteinuria (≥ 2+ on urine dipstick)
* Patient with congenital bleeding diathesis, acquired coagulopathy or under full dose of anticoagulants.
* Patient is currently receiving strong inducers or inhibitors of CYP3A4/5 or medication with narrow therapeutic window that are predominantly metabolized through CYP3A4/5 and cannot be discontinued 7 days prior to start of study treatment.
* Known presence of cerebral metastases unless at least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment and clinically stable central nervous system tumor at the time of screening.
* Patient is currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed.
* Patient is currently receiving or has received systemic corticosteroids or other chronic immunosuppressive therapy ≤ 2 weeks prior to starting study drug.
* Patients with advanced symptomatic, visceral spread, that are at risk of lifethreatening complications in the short term (including patients with massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver involvement).
* Patient has a known history of HIV infection (testing not mandatory).
* Patient has active untreated or uncontrolled fungal, bacterial or viral infection.
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, etc.).
* Participation in prior investigational studies within 30 days prior to randomization or within 5-half lives of the investigational product, whichever is longer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women (any menopausal status)
Enrollment: 41 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Efficacy in terms of PFS | Up to approximately 15 months.
  PFS is defined as time from randomization to progression of disease or death of any cause, whichever comes first. It will be assessed by imaging until progressive disease or start of next-line therapy.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 48 months.
  OS is defined as time from randomization to death of any cause.
Overall Response Rate (ORR) | Up to approximately 15 months.
  ORR is defined as the proportion of patients with best overall response of complete or partial response according to RECIST 1.1.
Clinical Benefit Rate (CBR) | Up to approximately 15 months
  CBR is defined as the proportion of patients with best overall response of complete or partial response or stable disease lasting 24 weeks or more according to RECIST 1.1.
Time To Response (TTR) | Up to approximately 15 months.
  TTR is defined as time from randomization to first occurrence of any response (complete or partial) according to RECIST 1.1.
Number of participants with Adverse Events | Until 30 days after end of treatment, up to approximately 16 months.
  Type, frequency and severity (according to CTCAE v4.03) of adverse events
Time to deterioration of ECOG performance status | Until 30 days after end of treatment, up to approximately 16 months
  Time to deterioration of ECOG performance status by at least one point from baseline.
Tolerability of treatment | Until 30 days after end of treatment, up to approximately 16 months.
  By-patient listings of safety laboratory (hemoglobin, platelets, white blood cells with differentials, international normalized ratio , serum creatinine, bilirubin, Alanine-Aminotransferase (ALT) and Aspartate-Aminotransferase (AST)).
corrected QT interval (QTc) time | Until 30 days after end of treatment, up to approximately 16 months.
  By-patient listings of cardiac monitoring.
Health-related quality of life (QoL) | Up to 36 months.
  Health-related QoL will be assessed with the EORTC Quality of life questionnaire (QLQ) QLQ-C30.
Side effects of treatment | Up to 36 months.
  One question on treatment burden
Time spent on treatment | Up to 36 months
  Burden by treatment will be assessed with 4 questions on time spent on treatment

OTHER OUTCOMES:
Symptomatic PFS (sPFS) | Up to approximately 15 months.
  sPFS is defined as time from randomization until symptomatic deterioration (new or worsening of persisting symptoms) or death as per local investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Decker, Prof., Principal Investigator — Gemeinschaftspraxis für Hämatologie und Onkologie
Locations (27):
- Germany (27):
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Ravensburg, Baden-Wurttemberg
  - Uniklinik RWTH Aachen, Gynäkologie und Geburtsmedizin, Aachen
  - Klinikum Mittelbaden Baden-Baden Balg, Baden-Baden
  - Gynäkologisches Zentrum Bonn, Bonn
  - St.-Johannes-Hospital Gynäkologie und Geburtshilfe, Dortmund
  - BAG / Onkologische Gemeinschaftspraxis, Dresden
  - Universitätsklinikum Essen, Essen
  - Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau
  - Überörtliche Berufsausübungsgemeinschaft MVZ Onkologische Kooperation Harz, Goslar
  - Gemeinschaftspraxis für Innere Medizin, Hämatologie, Onkologie, Gastroenterologie, Halle
  - OncoResearch Lerchenfeld GmbH, Hamburg
  - Onkologische Schwerpunktpraxis, Heidelberg
  - IDGGQ GbR, Kaiserslautern
  - Hämato-Onkologisches Zentrum Kassel MVZ GmbH, Kassel
  - Praxis Dr. med. Bettina Peuser, Leipzig
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Mühlheim
  - Hämatologisch-onkologische Gemeinschaftspraxis, Münster
  - Praxis Dr. med. Jens Uhlig, Naunhof
  - Klinikum Neumarkt, Neumarkt
  - Onkologie Offenburg, Offenburg
  - Praxis und Tagesklinik für Onkologie und Hämatologie, Recklinghausen
  - Tumorzentrum und Hausarztpraxis Rötha Leipziger-Land, Rötha
  - Schwerpunktpraxis für Hämatologie und Internistische Onkologie, Gastroenterologie, Singen
  - Onkologische Schwerpunktpraxis, Speyer
  - g.SUND Gynäkologie Kompetenzzentrum Stralsund, Stralsund
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Westerstede

IPD SHARING:
Plan to Share IPD: No